CLINICAL TRIAL: NCT01096134
Title: Mother - Daughter Initiative (MDI) in Cervical Cancer Prevention
Acronym: MDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Sharon Kibwana, Senior Program Officer, Jhpiego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 36448
Record Dates: First submitted 2010-03-23; First posted 2010-03-30 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Papillomavirus Vaccines; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HPV Vaccine (Experimental): Eligible girls were offered 3 doses of the HPV vaccine
  Interventions: Biological: HPV Vaccine (Gardasil)

INTERVENTIONS:
Biological: HPV Vaccine (Gardasil) — HPV Vaccine Administration: According to the CDC, Gardasil should be delivered through a series of three intra-muscular injections over a six-month period. The second and third doses should be given two and six months after the first dose. The vaccine can be administered at the same visit as other age-appropriate vaccines, such as Tdap, Td, MCV4, influenza, and hepatitis B vaccines. Providers should consider a 15-minute waiting period for vaccine recipients following vaccination.
  FDA's Approval of Gardasil (June 8, 2006) lists the following information on product Formulation: Each 0.5 mL dose of the vaccine contains:
  20 mcg of HPV 6 L1 protein 40 mcg of HPV 11 L1 protein 40 mcg of HPV 16 L1 protein 20 mcg of HPV 18 L1 protein 225 mcg aluminum (as amorphous aluminum hydroxyphosphate sulfate adjuvant) 9.56 mg of sodium chloride 0.78 mg of L-histidine 50 mcg of polysorbate 80 35 mcg of sodium borate water for injection

SUMMARY:
The Mother-Daughter Initiative (MDI) will test the feasibility and acceptability of a strategy to deliver comprehensive cervical cancer prevention services in Thailand and the Philippines by integrating the HPV vaccine for girls ages 9-13 into already successful screening and treatment programs for mothers.

ELIGIBILITY:
Inclusion Criteria:

* Age 9-13 at first HPV vaccine dose
* Mother/legal guardian and daughter are both interested and willing to have the girl receive the HPV vaccine
* Mother/legal guardian and daughter both indicate that they would be able to return to clinic for the three vaccine doses

Exclusion Criteria:

* Girls with a known history of any allergies or severe reaction to any vaccines, food or medicine
* Pregnant adolescents will be excluded. If a girl becomes pregnant after the first dose is administered, she will not be provided with the second or third dose
* Girls with moderate or severe illnesses will be asked to postpone vaccination eg. Pneumonia.
* Girls with a weakened immune system, cancer, leukemia, AIDS or other immune system problems
* Girls with a bleeding disorder or currently taking anticoagulants
* Girls that have received any other vaccinations in the past 4 weeks
* Girls currently on steroids, such as cortisone, prednisone, or anti-cancer drug.

Ages: 9 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8000 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Determine the population coverage of HPV vaccination of girls aged 9-13 offered within the context of cervical cancer screening and treatment of mothers | 18 months
  The aim of the study to assess whether we can fully vaccinate (all 3 doses),50% of girls aged 9 -13 in the participating districts, in an 18-month period. This corresponds to 4000 girls in Thailand and 4000 in Phillipines. The study will seek to undertand if this level of population coverage (50%), can be achieved through encouraging women that recive cervical cancer screening to bring in their daughters or relatives for vaccination.

SECONDARY OUTCOMES:
Assess mothers' acceptability of having their daughters receive the full course of HPV vaccine after mothers receive screening and treatment services for cervical pre-cancer | 1 year
  Data on mothers knowledge of the vaccine, and intention to have their daughters vaccinated will be collected for a period of 1 year (or when the target number of 700 women/guardians is reached, whatever comes first).
  Data will be collected on:
  * Proportion of women with daughters who intend to vaccinate their daughters.
  * Proportion of daughters of screened mothers who return to receive the vaccine.
  * Proportion of girls who receive the first vaccine dose and are brought to the facility by a guardian/mother who did NOT recieve cervical cancer screening
Inform future programs that aim to introduce the HPV vaccine in the context of secondary screening for cervical cancer by determining the factors related to screened women bringing daughters for HPV vaccination and the costs of vaccine introduction | 2 years
  Programmatic data will be collected for the duration of the project, including but not limited to:
  * Cost required to implement the program
  * Logistics required to ensure supply and appropriate maintenance of vaccine
  * Human resources required to effectively adminster the vaccine as part of routine services.
  * Key communication and outreach messages that effectively educate the community

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Llave, MD, Principal Investigator — Cancer Institute Foundation, Phillipines; Kobchitt Limpaphayom, MD, Principal Investigator — Chulalongkorn University, Thailand; Enriquito Lu, MD, MPH, Principal Investigator — Jhpiego
Locations (10):
- Philippines (3):
  - Minglanilla, Cebu
  - Los Banos, Quezon
  - Pagbilao Health Center, Quezon
- Thailand (7):
  - Health promotion Clinic Number 11, Nakhon Si Thammarat, Nakisron
  - Ban Pak Poon Health Center, Nakhon Si Thammarat, Nakornsri
  - Maharat Nakhonsithammarat Primary Care Unit, Nakhon Si Thammarat, Nakornsri
  - Pak-Panung District Health Center, Nakhon Si Thammarat, Nakornsri
  - Ban Yuanlae District Health Center, Ban Phon Ko
  - Ban Mai Daeng, Nakhon Si Thammarat, Nakornsri
  - Ban Pai Ta Health Center, Nakhon Si Thammarat, Nakornsri